CLINICAL TRIAL: NCT06816459
Title: Sensory Evaluation of Cigarettes Claiming Removal of Menthol as a Characterizing Flavor
Brief Title: Sensory Tests of Cigarettes for Identification of Flavors in Current Daily Smoking Adults
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: I-3571524; NCI-2025-00202 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3571524 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Cigarette Smoking-Related Carcinoma

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are blinded to brand and condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Block Alpha (block alpha cigarette tests) (Experimental): Participants complete 3 testing sessions, each session lasting 1 to 2 hours and each session at least 48 hours apart but no more than 1 week apart. Participants undergo the B-SIT during session 1, a block alpha cigarette smell test with a total of 16 cigarette products during session 2 and a block alpha cigarette taste test with a set of 3 cigarettes during session 3. Testing sessions are completed in the absence of illness or unacceptable toxicity.
  Interventions: Other: Cigarette smell test; Other: Cigarette Taste Test; Other: Study questionnaires
- Block Beta (block beta cigarette tests) (Experimental): Participants complete 3 testing sessions, each session lasting 1 to 2 hours and each session at least 48 hours apart but no more than 1 week apart. Participants undergo the B-SIT during session 1, a block beta cigarette smell test with a total of 16 cigarette products during session 2 and a block beta cigarette taste test with a set of 3 cigarettes during session 3. Testing sessions are completed in the absence of illness or unacceptable toxicity.
  Interventions: Other: Cigarette smell test; Other: Cigarette Taste Test; Other: Study questionnaires

INTERVENTIONS:
Other: Cigarette smell test — Undergo cigarette smell test of 16 cigarettes in vials, then rate the overall smell on a 5 pt scale (not at all, a little noticeable, noticeable, clearly/very noticeable , do not know what this is).
Other: Cigarette Taste Test — Participants will be present 3 vials , each containing a cigarette and sample in order specified on label, then complete a coolness measure on a 0-100 visual analog scale.
  Other Names: Taste Test
Other: Study questionnaires — Sensory questionnaires will be administered using a web based application

SUMMARY:
This clinical trial tests how well current daily smoking adults can identify flavors of cigarettes. Menthol cigarettes account for 31 percent of cigarettes sold in the United States. Flavors such as menthol play an important role in the start and continued use of tobacco products. Two ways users experience flavor is through smell and taste. Menthol has cooling and numbing properties that can increase perceptions of smoothness and reduce the perceived harshness of smoke. Menthol adds a taste and aroma commonly described as "minty". The effect of menthol flavoring on smoking behavior has been studied. Use of menthol cigarettes has been associated with greater nicotine dependence and is associated with both fewer quit attempts and lower odds of quit success. In 2022, the Food and Drug Administration proposed to restrict the use of menthol as a flavor in cigarettes. Menthol has already been banned in Canada, the United Kingdom and the European Union. In late 2022, a restriction on all flavored tobacco products went into effect in California (CA), prompting the tobacco industry to introduce substitute products that did not contain menthol. It is important to find out whether New York (NY) adult smokers who smoke menthol cigarettes can identify and characterize flavors in the same cigarette brand as sold in NY versus CA following the ban of menthol cigarettes in 2022.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To convene a consumer panel of adult smokers in New York state (N=24) to assess the smelling properties of a sample of cigarette products sold in the New York and California markets to identify any characterizing flavors.

EXPLORATORY OBJECTIVE:

I. To collate consumer-test findings, highlighting quantitative analysis of any characterizing flavors identified, as well as any qualitative insights from the panel about specific products.

OUTLINE: Participants are randomized to 1 of 2 blocks.

BLOCK ALPHA: Participants complete 3 testing sessions, each session lasting 1 to 2 hours and each session at least 48 hours apart but no more than 1 week apart. Participants undergo the Brief Smell Identification Test (B-SIT) during session 1, a block alpha cigarette smell test with a total of 16 cigarette products during session 2 and a block alpha cigarette taste test with a set of 3 cigarettes during session 3. Testing sessions are completed in the absence of illness or unacceptable toxicity.

BLOCK BETA: Participants complete 3 testing sessions, each session lasting 1 to 2 hours and each session at least 48 hours apart but no more than 1 week apart. Participants undergo the B-SIT during session 1, a block beta cigarette smell test with a total of 16 cigarette products during session 2 and a block beta cigarette taste test with a set of 3 cigarettes during session 3. Testing sessions are completed in the absence of illness or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-55 years old
* Current daily smoker of factory-made menthol cigarettes
* General good health (assessed by self-rated health item)
* Completion of Brief Smell Identification Test (B-SIT) with no identification of deficits

Exclusion Criteria:

* Daily concurrent use of other tobacco products (e.g., e-cigarettes, cigars, smokeless tobacco)
* Known allergies to mint (peppermint, spearmint), menthol
* Self-reported olfactory or taste deficits
* Pregnant or nursing participants, as indicated by self-report
* History of medications known to interfere with sense of smell
* Positive diagnosis of coronavirus 2019 (COVID-19) within 10 days of enrollment
* Current upper respiratory infection or sinus congestion (e.g., cold, flu, seasonal allergies) (by self report)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Menthol smell presence | Up to 1 year
  Will evaluate ratings of menthol smell presence (0-5 scale). Data will be analyzed under the generalized linear model approach, a flexible regression-based approach that allows for different distributional assumptions of the dependent variable, and for different link functions to describe the relationship between the independent and dependent variable. These models utilize maximum likelihood (iteratively reweighted least squares) estimation. The generalized estimating equation extension allows for modeling of sample-averaged repeated measures within individuals.
Mint-like smell | Up to 1 year
  Will evaluate ratings of mint-like smell (0-4 scale). Data will be analyzed under the generalized linear model approach, a flexible regression-based approach that allows for different distributional assumptions of the dependent variable, and for different link functions to describe the relationship between the independent and dependent variable. These models utilize maximum likelihood (iteratively reweighted least squares) estimation. The generalized estimating equation extension allows for modeling of sample-averaged repeated measures within individuals.
Cooling sensation during taste test | Up to 1 year
  Will be assessed using a self-rated coolness measure on a 0-100 visual analog scale. Data will be analyzed under the generalized linear model approach, a flexible regression-based approach that allows for different distributional assumptions of the dependent variable, and for different link functions to describe the relationship between the independent and dependent variable. These models utilize maximum likelihood (iteratively reweighted least squares) estimation. The generalized estimating equation extension allows for modeling of sample-averaged repeated measures within individuals.

SECONDARY OUTCOMES:
California (CA) version of the test brand cigarette | Up to 1 year
  Will evaluate proportion correctly identifying the CA version of the test brand cigarette.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J O'Connor, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States